CLINICAL TRIAL: NCT01271569
Title: A Phase 1,Open, Dose-escalation Study to Assess the Efficacy and Safety of Fospropofol Disodium Injection in Healthy Volunteers
Brief Title: A Study to Assess the Efficacy and Safety of Fospropofol Disodium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: West China Hospital, Sichuan University, West China Hospital, Sichuan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFDA2009L09746; 2009L09746 (Other: the State Food and Drug Administration in China)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2010-03

CONDITIONS: Drug Safety
MeSH Terms: interventions — fospropofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- In the treatment arm (Other)
  Interventions: Drug: Fospropofol disodium

INTERVENTIONS:
Drug: Fospropofol disodium — Fospropofol disodium： 0.5g

SUMMARY:
The aim of this study was to evaluate the pharmacodynamics, safety, and tolerability of Fospropofol disodium up to a dose producing maximal hypnotic effect as defined by electroencephalogramderived assessment (Bispectral Index [BIS]) and to compare the dynamic properties of PropofolF to those of Propofol.

DETAILED DESCRIPTION:
After local ethics committee (West China Hospital, Sichuan University, Chengdu, China) approval and written informed consent were obtained, 80 healthy volunteers (40 males and 40 females) aged between 18 and 45 yr were included. For 1 week before the study, subjects were to follow a diet with limited amounts of alcohol and caffeine. Ingestion of caffeine, alcohol, products containing aspartame (aspartame may increase formate concentrations), or use of paracetamol within 24 h before study drug administration resulted in ineligibility. Exclusion criteria included hypersensitivity to any anesthetic; known or suspected serious disorders and/or significant dysfunction; an abnormal, clinically significant ECG finding; participation in an investigational drug study within the previous month; known or suspected pregnancy; anatomical malformations expected to produce a difficult intubation and known or suspected history or family history of malignant hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* After local ethics committee (West China Hospital, Sichuan University, Chengdu, China) approval and written informed consent were obtained, 80 healthy volunteers (40 males and 40 females) aged between 18 and 45 yr were included. For 1 week before the study, subjects were to follow a diet with limited amounts of alcohol and caffeine.

Exclusion Criteria:

* Exclusion criteria included hypersensitivity to any anesthetic; known or suspected serious disorders and/or significant dysfunction; an abnormal, clinically significant ECG finding; participation in an investigational drug study within the previous month; known or suspected pregnancy; anatomical malformations expected to produce a difficult intubation and known or suspected history or family history of malignant hyperthermia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
BIS | 2hr after administration

SECONDARY OUTCOMES:
Modified OAA/S Score | 2hr after administration

CONTACTS AND LOCATIONS:
Overall Officials: Jin Liu, MD, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China